CLINICAL TRIAL: NCT00444197
Title: Community-Based Violence Prevention for High-Risk Youth
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R40MC00174-01
Record Dates: First submitted 2007-03-05; First posted 2007-03-07 (Estimated); Last update posted 2007-03-07 (Estimated); Status verified 2007-03

CONDITIONS: Fighting Behavior; Aggression
MeSH Terms: conditions — Aggression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Mentoring and violence prevention curriculum with parental monitoring

SUMMARY:
Study Aims: 1) Assess the receptiveness of youth and families to injury prevention interventions initiated from the emergency department; 2) In a sample of high risk youth presenting to the ED with interpersonal assault injuries, determine the effectiveness of a home-based family intervention with community linkage compared to a control group.

DETAILED DESCRIPTION:
The leading causes of death among U.S. children and adolescents are due to injuries. In the US, homicide is the third leading cause of death for 10-14 year olds and second leading cause of death for those 15-19 years. For African-Americans, homicide is the leading cause of death for males and females ages 15-34. Findings from our city-wide surveillance of adolescent injuries have found that for every death due to injury in youth, there were 8 hospitalizations and 102 ED visits. Non-fatal injuries represent significant morbidity and may be a sentinel event and opportunity for prevention.

Assault-injured patients age 9-15 and their families seen in the ED or hospitalized will be recruited into the study. Whenever possible, families will be recruited while they are still in the hospital, others will be contacted by phone. We will randomize families to an intervention group consisting of home visits involving a four session parental monitoring curriculum for parents and a 6-8 session mentoring and problem solving curriculum for youth occurring over 2-6 months. Both intervention and control groups will receive community referrals to needed services. Interview assessments of parents and youth will occur in person at baseline and 6 months, and by phone at 12 and 18 months after recruitment. Assessments will include face to face and Walkman questioning, and phone questioning with DigitGrabber touch tone response. The parent and youth assessments will include detail on cause of injury, past experience risk factors, protective factors, perceived risk and self-efficacy. Medical chart abstraction will be performed and aggregate data will be obtained from the police department about the number of youth in the intervention and control groups that have had contact with the police. We intend to recruit up to 400 families over 2-3 years in order to achieve follow-up with at least 198 families. Human Subjects: Male and female adolescents 9-15 years of age and their parents who are residents of the Washington Metropolitan area will be eligible for participation. Written parental consent and youth assent will be obtained. There are no physical risks. Potential risks include unintentional uses of the information gathered including disclosure of information that may be potentially legally incriminating. All efforts will be made to protect participant confidentiality. If information is revealed that places someone in immediate danger, disclosure may be necessary which is explained in the consent form. There are potential benefits including facilitated referral for therapeutic community-based intervention, access to an intervention of demonstrated effectiveness without cost, and cash incentives. In addition, they will contribute to knowledge about youth injury in the community.

ELIGIBILITY:
Inclusion Criteria:

* adolescents age 9-15 presenting to a large urban children's hospital or university hospital
* residence in the metropolitan area
* emergency department presentation with an interpersonal assault injuries (E960, 961-966, 968-969) excluding sexual assault, child abuse, sibling fights, or legal intervention
* mental and physical ability of parent and child to participate in the intervention and assessments.

Exclusion Criteria:

* sexual assault, child abuse, sibling fights, or legal intervention
* non English speaking

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 198
Dates: Start 2001-08; Study Completion 2006-01

PRIMARY OUTCOMES:
Fighting behavior
Weapon carrying
Aggression
Misdemeanors

SECONDARY OUTCOMES:
Attitudes About Violence
Self Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Tina L Cheng, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins University, Baltimore, Maryland

REFERENCES:
- [Derived] Cheng TL, Haynie D, Brenner R, Wright JL, Chung SE, Simons-Morton B. Effectiveness of a mentor-implemented, violence prevention intervention for assault-injured youths presenting to the emergency department: results of a randomized trial. Pediatrics. 2008 Nov;122(5):938-46. doi: 10.1542/peds.2007-2096. PMID 18977971